CLINICAL TRIAL: NCT05801809
Title: Understanding the Effects of Non-invasive Transauricular Vagus Nerve Stimulation (taVNS) on Neural Networks and Autonomic Nervous System: a Randomized Double-blind Sham-control Mechanistic Trial in Healthy Participants
Brief Title: Understanding the Effects of Transauricular Vagus Nerve Stimulation on Neural Networks and Autonomic Nervous System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Director of Spaulding Neuromodulation Center, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2022P003200
Record Dates: First submitted 2023-02-27; First posted 2023-04-06 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: vagal nerve stimulation; healthy subjects; biomarkers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active taVNS (Experimental): TaVNS will be administered by an earset, with conductive eartips placed on the auricular concha of the ears, connected to a stimulator, and during active stimulation, we stimulate both the cymba conchae and external auditory canal of both left and right ears with the following parameters: 30Hz, 200-250 us, and with adjustable intensity for 60 min.
  Interventions: Device: Transauricular vagus nerve stimulation (taVNS)
- Sham taVNS (Sham Comparator): Sham condition will have the same device, with an earset, and conductive eartips placed in the same location of the active stimulation; however during 60 min there will be no current and the device will be turned off.
  Interventions: Device: Transauricular vagus nerve stimulation (taVNS)

INTERVENTIONS:
Device: Transauricular vagus nerve stimulation (taVNS) — Transauricular vagus nerve stimulation (taVNS) is a simple technique in which small surface electrodes are placed over the skin of the ear that are thought to be innervated by the auricular branch of the vagus nerve (ABVN).

SUMMARY:
This trial aims to perform an exploratory, mechanistic, randomized double-blind sham-control trial in healthy participants to assess the physiologic effects of a single 60 minutes session of bilateral taVNS, on neural networks and autonomic function.

DETAILED DESCRIPTION:
Several studies have shown promising results of taVNS to treat various disorders such as depression, anxiety, Alzheimer's disease, headache, obesity, and diabetes. However, no mechanistic studies have investigated the taVNS neural network and autonomic nervous system effects of this technique. Therefore, we aim to assess how taVNS can affect EEG metrics and HRV and assess its safety. Also, we aim to evaluate predictors that can influence the response to taVNS, so understanding the variables associated with response to taVNS can help the design of future clinical trials to maximize the effects of this intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to participate in the study.
2. Subject is older than 18 years.
3. Subjects should be naive to the stimulation (taVNS)

Exclusion Criteria:

1. Pregnancy.
2. Subjects who have had a neuropsychiatric or a cardiac disorder diagnosis and have received treatment and chronic medication in the past six months, or who have functional deficits as a result.
3. History of alcohol or drug abuse within the past 6 months as self-reported.
4. Presence of the following contraindication to transauricular vagus nerve stimulation

   1. Ferromagnetic metal in the head and in the cranium (e.g., plates or pins, bullets, shrapnel)
   2. Implanted cranial electronic medical devices (e.g., cochlear implants)
   3. Implanted cardiac devices (e.g., pacemaker)
5. Unstable medical conditions (e.g. uncontrolled diabetes, uncompensated cardiac issues, heart failure, or chronic obstructive pulmonary disease).
6. Uncontrolled epilepsy, as defined by previous clinical seizures in the past 3 months in patients with treatment for epilepsy.
7. Suffering from severe depression (as defined by a score of >30 in the Beck Depression Inventory).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2026-03-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital/Harvard Medical School
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active taVNS | Sham taVNS
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active taVNS | Sham taVNS | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (68.2) | 40.8 (17.8) | 41.3 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 14 | 11 | 25
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Resting-state Electroencephalogram (EEG)
Description: Resting-state EEG was recorded using a 64-channel high-density EGI system (Electrical Geodesics, Inc., Eugene, USA) under the eyes closed condition. Data was filtered into standard frequency bands using short-time Fourier transformation (STFT): delta (0.5-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), and gamma (30-80 Hz).
  Frontal asymmetry was computed as the difference in power between homologous left and right frontal electrodes (e.g., F3-F4) in the alpha band.
Time Frame: Change from baseline to 60 minutes post-intervention.
Measure: Mean (Standard Deviation); unit: Difference in alpha asymmetry (µV²).
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 21 | 22
Difference in alpha asymmetry (µV²). | 0.016 (0.012) | -0.025 (0.016)

2. Primary Outcome: Conditioned Pain Modulation (CPM) Response - Change in Pain Ratings on the Pain-6 Scale (0-10)
Description: Pain intensity was measured using the Numeric Pain Scale (NPS; 0 = no pain, 10 = worst pain). Higher scores indicate worse pain. A "pain-6 temperature" was first identified (temperature that elicits NPS = 6).
  Test stimulus: Pain-6 temperature applied for 30s; participants rated pain at 10, 20, and 30s. The test-stimulus score is the average of the three NPS ratings.
  Conditioned stimulus: After 5 minutes, the left hand was immersed in 10-12°C water for 30s while the same pain-6 temperature was applied again. Pain was rated the same way, and the conditioned-stimulus score is the average of the three NPS ratings.
  CPM calculation = (test-stimulus average) - (conditioned-stimulus average). Positive values = better endogenous pain inhibition; negative values = worse.
Time Frame: Change from baseline to 60 minutes post-taVNS.
Measure: Mean (Standard Deviation); unit: Unit on a scale (NPS 0-10)
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 22 | 19
Unit on a scale (NPS 0-10) | 0.34 (0.60) | -0.53 (1.14)

3. Secondary Outcome: Heart Rate Variability (HRV)
Description: HRV from ECG on non-dominant hand. High-frequency HRV calculated from 5-min resting recordings; higher values indicate greater parasympathetic activity. Post-stimulation values (60 min) were analyzed.
Time Frame: Post-intervention (after 60 minutes of taVNS)
Measure: Mean (Standard Deviation); unit: ms²
Arm/Group | Active taVNS | Sham taVNS
Number analyzed (Participants) | 22 | 22
ms² | 0.6 (0.3) | 0.1 (0.2)

ADVERSE EVENTS:
Time Frame: Side effects were assessed on the same day, immediately after the stimulation.
Description: No serious or unforeseen adverse events were documented. Only one participant in the active group reported transient tingling behind their left ear at the onset of stimulation, dissipating within the subsequent five minutes.
Arm/Group | Active taVNS | Sham taVNS
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 1/22 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active taVNS (N=22) | Sham taVNS (N=22)
Expected side effect (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Transient tingling behind their left

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT05801809/Prot_SAP_002.pdf